CLINICAL TRIAL: NCT02488265
Title: Randomized Controlled Trial Protocol: Balance Training With Rhythmical Cues to Improve and Maintain Balance Control in Parkinson's Disease
Brief Title: Protocol: Balance Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tamine Capato 02
Record Dates: First submitted 2015-05-21; First posted 2015-07-02 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson´s disease; Physicaltherapy; Postural Balance; Gait; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motor training (Experimental): Balance training, Screening to prevent falls
  Interventions: Other: Balance Training; Other: Screening to prevent falls
- Balance RhytmicalTraining (Experimental): Balance training, Screening to prevent falls
  Interventions: Other: Balance Training; Other: Screening to prevent falls

INTERVENTIONS:
Other: Balance Training — Balance training with rhythmical (BRT), is a motor program to improve balance associated with rhythmical auditory cues (RACs).
Other: Screening to prevent falls — Questionary to Scheduled screening falls and progression in training will be used to indicate the capacity to continue to progress.

SUMMARY:
Postural instability is a particularly incapacitating disorder, where loss of motor independence by Parkinson´s Disease (PD) patients marks a significant stage of disease onset. Evidence suggests that deficits in automatic motor control, sensory integration and attention are associated with lack of balance in PD. Physiotherapy, together with medication, plays an important role in the treatment of this state, although no consensus has been reached on the best treatment modality. The aim of this randomized controlled trial protocol is to evaluate the effects of balance training with rhythmical (BRT), which is a motor program to improve balance associated with rhythmical auditory cues (RACs)

DETAILED DESCRIPTION:
A total of 150 PD patients at H&Y stages II-III and asymptomatic for depression and dementia are enrolled in a single-blind randomized study. Randomization is achieved via a computer-generated random-sequence table. All patients should also present a fall history.They will be assigned into one of three groups, and their balance and gait will be assessed before and after 10 training sessions, and after 4 and 30 weeks subsequent to the end of the training. Balance will be assess by Mini BESTest (MBESTest), BERG Test (BBS) and Postural Stress Test (PST). Gait will be evaluate by the Timed Up and Go test (TUG). Independence in Activities of Daily Living (ADLs) will be assess through interviews; and UPDRS, through motor performance. The BRT group received a motor program to improve balance associated with RACs, the MT group performed motor training with the same aims as those in the BRT group but without RACs, and the control group (CG) was trained only in orientations. The exercise program specific to balance is of 5 weeks' duration with two sessions per week, 45 minutes each, and consists of general physiotherapy exercises. Each session is divided into five warm-up minutes-30 minutes for the main part and 10 minutes for the cool down. The training progresses and intensifies each week depending on the individual's performance. The subjects should be able to execute 10 repetitions of the exercise sequences correctly to progress to the next movement.

The training progressed and increased in intensity on each week. On the first week, before the training, each exercise was explained and demonstrated by the physiotherapist, who demanded special attention on the most difficult aspects of movement execution. The subjects performed 05 repetitions (5 RM) of each exercise.

On the first phase the patients may present some mistakes and might need specific information to correct the movement that is on execution. The exercises will be repeat in the next sessions in order to consolidate learning. The subjects must have been capable of associating the corrections to the exercises that will proposs on the first week. In each group repetition, for both groups, the physiotherapist will use a verbal command before each movement change, anticipating it and requesting attention to the most difficult ones. Only the GBRT will be oriented to focus on the rhythmical auditory cues. On the second week, the subjects will perform a series of 10 repetitions (10 RM) and on the third week, 2 series of 10 repetitions (20RM). On the fourth week, subjects must have been able to execute 20RM of the exercise sequences with an increase in speed.

ELIGIBILITY:
Inclusion Criteria:

* All of the subjects will be diagnosed by neurologists from the Movement Disorders Ambulatory Clinic of the University of São Paulo Faculty of Medicine Clinics Hospital, according to the UK Brain Bank criteria [36] and should be at H&Y classification stage II or III, with a Mini Mental Status Examination (MMSE) [37] score of above 24.
* All patients should also present fall history.
* They should have the capacity to ambulate independently indoors without aid.

Exclusion Criteria:

* These are the presence of neurological, orthopedic or cardiopulmonary problems, an unstable medication regime, and an inability to understand or adhere to the protocol because of, for example, cognitive, auditory or visual problems.
* Patients receiving physical therapy training will also be excluded from the training.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Mini BESTest (MBESTest) | 30 weeks
  Clinical balance assessment tool that aims to target different balance control systems so that specific rehabilitation approaches can be designed for different balance deficits.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | 30 weeks
  Berg Balance Scale assesses the functional balance of patients with Parkinson´s disease. It is a clinic assessment of patient that evaluate the antecipatory postural adjustments and the performance of patient to stand up and sit down, turn on and step, among others situations.
UPDRS | 30 weeks
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a rating scale used to follow the longitudinal course of Parkinson's disease
Timed Up and Go test (TUG) | 30 weeks
  The Timed Up and Go test is a short, practical test by which gait and balance are tested
Push and Release Test | 30 weeks
  by which an unexpected, quick and firm jerk on the shoulder is given in a backward direction.It is a clinic assessment of patient that evaluate the compensatory postural adjustments
New Freezing of gait questonary (NFoG) | 30 weeks
  Questionay - measures of freezing of gait
Falls Efficacy Scale-International (FES-I) | 30 weeks
  The FES-I is a scale used to assessment the fear of falling.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PhD, Study Director — University of Sao Paulo; Tamine TC Capato, Master, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo Clinical Hospital, São Paulo, Brazil

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Capato TTC, de Vries NM, IntHout J, Ramjith J, Barbosa ER, Nonnekes J, Bloem BR. Multimodal Balance Training Supported by Rhythmic Auditory Stimuli in Parkinson Disease: Effects in Freezers and Nonfreezers. Phys Ther. 2020 Oct 30;100(11):2023-2034. doi: 10.1093/ptj/pzaa146. PMID 32737973
- [Derived] Capato TT, Tornai J, Avila P, Barbosa ER, Piemonte ME. Randomized controlled trial protocol: balance training with rhythmical cues to improve and maintain balance control in Parkinson's disease. BMC Neurol. 2015 Sep 7;15:162. doi: 10.1186/s12883-015-0418-x. PMID 26347052